CLINICAL TRIAL: NCT03566875
Title: Etude Clinique, Monocentrique, Prospective, randomisée et contrôlés de l'Arthoplastie Totale de Genou Avec le système Robotique MAKO™ Par Rapport à l'Arthroplastie Totale de Genou Conventionnelle Par Ancillaire mécanique
Brief Title: Total Knee Arthroplasty Robot Assisted With MAKO™ Robotic System Compared to the Conventional Total Knee Arthroplasty by Mechanical Ancillary
Acronym: TKA-MAKO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Clinical Investigation Centre for Innovative Technology Network (Network); Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 38RC17.373
Record Dates: First submitted 2018-06-12; First posted 2018-06-25 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Total Knee Arthroplasty
Keywords: TKA robot assisted with the Stryker's MAKO™ system; surgery precision
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total knee arthroplasty with the Stryker's MAKO™ system (Experimental): The total knee arthroplasty is performed with Stryker's MAKO™ robotic system. It allows to place precisely the prosthetic implants.
  Interventions: Procedure: Total knee arthroplasty with the Stryker's MAKO™ system
- Total knee arthroplasty with mechanical ancillary (Active Comparator): The total knee arthroplasty is performed using a mechanical ancillary. It's the conventional method.
  Interventions: Procedure: Total knee arthroplasty with mechanical ancillary

INTERVENTIONS:
Procedure: Total knee arthroplasty with the Stryker's MAKO™ system — The robot assisted surgery is performed using the Stryker's MAKO™ system. The precision with this system is very accurate. It should help the surgeon to improve the positioning accuracy of prosthetic implants compared to the conventional method.
  Arms: Total knee arthroplasty with the Stryker's MAKO™ system
Procedure: Total knee arthroplasty with mechanical ancillary — The arthroplasty is performed with the mechanical ancillary refering to the the conventional method.
  Arms: Total knee arthroplasty with mechanical ancillary

SUMMARY:
For the total knee arthrorplasty (TKA), the placement of a prosthesis is delicate and the correct positioning of the implants determines the result of the surgery.

Navigation has improved surgical accuracy but remains inadequate with nearly 20% malposition. In the early 2010s, robot-assisted surgery solutions were born. Amongst its offers, Stryker's MAKO™ system appears to be the most advanced and developed due to its precision and its flexibility of use during surgery.

In this study, the investigators evaluate the placement of the total knee prosthesis with the MAKO™ system compared to the placement of the total knee prosthesis with a conventional mechanical system for TKA

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Patient who must have a total prosthetic knee surgery at CHUGA with the useful indications : painful and disabling knee joint disease: traumatic arthritis or avascular necrosis, rheumatoid arthritis or post-traumatic arthritis, post-traumatic loss of the configuration and function of the knee joint, moderate deformities in varus, or valgus or flexion in ligamentous structures can find a function and a fracture of the distal femur and / or proximal tibia that can not be stabilized by standard fracture management techniques.
* Social security affiliates or beneficiaries of a scheme

Exclusion Criteria:

* refusal of consent,
* patient with a contraindication to prosthetic knee surgery:
* any active or suspected latent infection in or around the knee joint,
* remote foci of infection that can cause haematogenous spread on the implant site,
* any mental or neuromuscular disorder that would create an unacceptable risk of instability of the prosthesis,
* failure of prosthesis fixation or complications in postoperative care,
* a bone stock compromised by a disease,
* infection or anterior prosthetic implantation that can not provide adequate support and / or satisfactory fixation to the prosthesis,
* skeletal immaturity,
* severe instability of the knee joint secondary to the lack of integrity and function of the collateral ligament,
* woman of childbearing age,
* patient during the exclusion period of another study,
* patient referred in Articles L1121-5 to L1121-8 of the Public Health Code

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-04-23 (Actual); Primary Completion 2020-09-23 (Estimated); Study Completion 2020-09-23 (Estimated)

PRIMARY OUTCOMES:
Difference between the actual HKA angle obtained postoperatively and the planned HKA angle preoperatively. | 26 months
  HKA (Hip-Knee-Ankle). Angles in degrees are obtained from preoperative 3D scanner and postoperative 3D scanner on day 7.

SECONDARY OUTCOMES:
To compare the mechanical axis between the conventional surgery group and the MAKO™ assisted surgery group. | 26 months
  Mechanical axis (in degree) evaluated from the post-operative 3D computed tomography on the day 7.
To compare, between the conventional surgery group and the MAKO™ assisted surgery group, the angles accuracy of inclination and rotation in the 3 planes of the space (frontal, sagittal and axial) to accomplish the preoperative planning. The accuracy | 26 months
  difference between the angles of inclination and rotation obtained postoperatively and the planned angles preoperatively, in the 3 planes of the space. The angles, in degree, are evaluated from 3D preoperative scan and postoperative 3D scan.
To compare the operative time between the conventional surgery group and the MAKO™ assisted surgery group. | 26 months
  Duration (in minutes) between the time of the last stitch and the time of the first incision.
To evaluate the conversion rate in conventional method for patients in the MAKO™ assisted surgery group. | 26 months
  Conversion number to conventional method.
To compare the blood loss during the procedure between the conventional surgery group and the MAKO™ assisted surgery group. | 26 months
  Blood loss in liter according to the BRECHER formula (see Appendix E).
To compare between the conventional surgery group and the MAKO™ assisted surgery group the time needed to reach the hospital discharge criteria. | 26 months
  Duration (in days) between the date of the surgery and the date on which the patient can ascend the stairs on one floor and walk 100 meters with a cane.
To compare the functional results between the conventional surgery group and the MAKO™ assisted surgery group. | 26 months
  KSS, KOOS and EQ5D-3L scores at inclusion, then at 3 months, 6 months, and 1 year postoperatively.
To compare intraoperative complication rates between the conventional surgery group and the MAKO™ assisted surgery group. | 26 months
  Number of intraoperative complications. The complications are classified according to the following classification: light grade 1; moderate level 2; severe grade 3.
To compare the results of early (<1 months) and late (≥ 1 month) postoperative consultations between the conventional surgery group and the MAKO™-assisted surgery group. | 26 months
  Number of early (<1 month) and late (≥ 1 month) postoperative complications. Complications are classified according to the following classification: mild grade 1; moderate level 2; severe grade 3
To compare between the conventional surgery group and the MAKO™-assisted surgery group the operating times for surgical installation, bone preparation and implant placement. | 26 months
  1. for the surgical installation step: duration in minutes between the start of installation time (= end of anesthesia) and the time of first incision;
  2. for the bone preparation step: duration in minutes between the time of the first incision and the hour of end of extraction of the femoral sections;
  3. for the implant placement stage: duration in minutes between the start time of placement of the trial tibial implant and the time of the last stitch.

CONTACTS AND LOCATIONS:
Overall Officials: Régis Pailhé, PhD, Principal Investigator — Centre Hospitalier Universitaire Grenoble-Alpes
Locations (1):
- University Grenoble Hospital, Échirolles, France